CLINICAL TRIAL: NCT05212805
Title: Aerobic Training as Substrate for Neural Plastic Changes in Multiple Sclerosis: a Putative Disease-modifying Treatment?
Brief Title: Promoting Aerobic Training in Multiple Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Italiana Sclerosi Multipla (Other)
Collaborators: Universita degli Studi di Genova (Other); University Grenoble Alps (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARSEP
Record Dates: First submitted 2021-11-02; First posted 2022-01-28 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Multiple Sclerosis
Keywords: Aerobic exercise; Sports activity; Motor performance; Neural plasticity; Participation; Upper limb
MeSH Terms: conditions — Multiple Sclerosis | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic Exercise Promotion (Experimental): This group will be submitted to an aerobic exercise program combined with upper-limb motor training.
  Interventions: Behavioral: Aerobic exercise; Behavioral: Task-oriented upper-limb training; Behavioral: Sport events participation
- Control (Active Comparator): This group will be submitted to a standard motor rehabilitation. No aerobic nor sport activity will be delivered to the Control group.
  Interventions: Behavioral: Task-oriented upper-limb training

INTERVENTIONS:
Behavioral: Aerobic exercise — Interventions will be delivered through twenty supervised 40-minutes aerobic sessions (3 times a week). Patients will be trained on a bicycle ergometer (5-minute warm-up, 30 minute of intense training, 5-minute cool-down). Warm-up will be performed at the 30% of the maximal heart rate, while training will be performed at the 50-70% of the maximal heart rate as recommended by the general guidelines for aerobic exercise training specific for MS. Actual heart rate will be constantly monitored by a wearable heart rate monitor.
  Arms: Aerobic Exercise Promotion
Behavioral: Task-oriented upper-limb training — The training will consist in twenty 1-hour sessions (3 times a week) of exercises for neuromuscular control to improve proprioceptive sensibility, muscle strength, stability and coordination of the upper limbs, including unimanual and bimanual task-oriented exercises.
Behavioral: Sport events participation — A subgroup of participants will also be involved in events promoting sports activity including both aerobic and task-oriented exercises (e.g., water sports such as sailing, windsurfing, canoeing) in order to evaluate their potential role to increase adherence to training, participation and quality of life.
  Arms: Aerobic Exercise Promotion

SUMMARY:
Multiple sclerosis (MS) is a chronic neurological disease characterized by inflammation and degeneration within the central nervous system. Over the course of the disease, most patients with MS successively accumulate inflammatory lesions and axonal damage with an increasing degree of disability. Thus, pharmacological treatment options are currently adopted to limit inflammation and to decrease the relapse rate, or simply to alleviate symptoms. On the other hand, neurorehabilitation aims to maintain and possibly improve the residual capacities of neurological patients in order to preserve personal and social activities, constituting an important part of quality health care for MS patients. However, to date, there is no definite agreement on which specific exercise therapy program can be considered the most successful in improving activities and participation. Several studies suggest that a training based on voluntary movements produces greater improvements than a passive treatment. Aerobic exercise training has been also shown to have significant neurophysiological effects in different populations. Furtherly, sports activity may increase adherence and motivation, especially in a young population such as the MS community. However, feasibility of sports activity has not been investigated yet and, in general, the potential interest of these approaches for MS patients remains to determine.

This study aims at promoting physical activity in people with MS. Specific objectives are: (i) to evaluate the motor behavioral and neural changes induced by aerobic exercise combined with upper limb motor training based on task-oriented exercises; (ii) to assess the feasibility of leisure time physical activity (e.g. water sports activities) largely involving upper limb function.

Participants will receive task-oriented treatment, but only the experimental group will perform also aerobic training in order to evaluate the effect of aerobic exercise. Moreover, the role of sports activities will be preliminary investigated, by promoting the participation of the included patients to local or national events focusing on adapted aerobic sports specifically involving upper limb function (e.g., water sports such as sailing, windsurfing, canoeing). Clinical measures will be performed before and after interventions.

ELIGIBILITY:
Inclusion Criteria:

* Multiple sclerosis diagnosis according to McDonald criteria
* relapsing-remitting course
* absence of relapses in the last three months
* an Expanded Disability Status Score (EDSS) ≤ 4

Exclusion Criteria:

* steroid-use, psychiatric disorders or severe cognitive impairment
* acute cardio-respiratory diseases
* magnetic resonance imaging contraindications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2023-06-24 (Estimated); Study Completion 2023-12-25 (Estimated)

PRIMARY OUTCOMES:
Change in the 6 minute walk test (6mWT) performance | Baseline (T0), after 5 days of sports activity (Ti, if applicable), after 8 weeks (T1), after 16 weeks (T2)
  The 6mWT assesses distance walked over 6 minutes as a sub-maximal test of aerobic capacity/endurance

SECONDARY OUTCOMES:
Change in the Timed 25-Foot Walk test (T25FW) performance | Baseline (T0), after 5 days of sports activity (Ti, if applicable), after 8 weeks (T1), after 16 weeks (T2)
  The T25FW is a clinical tool that evaluates patients for quantitative mobility and leg function performance test in a timed, 25 foot walk
Change in the Nine Hole Peg Test (NHPT) performance | Baseline (T0), after 5 days of sports activity (Ti, if applicable), after 8 weeks (T1), after 16 weeks (T2)
  The NHPT is a standardized, quantitative assessment used to measure finger dexterity
Change in the Modified Fatigue Impact Scale (MFIS) score | Baseline (T0), after 5 days of sports activity (Ti, if applicable), after 8 weeks (T1), after 16 weeks (T2)
  The MFIS is a patient reported outcome on the effects of fatigue in terms of physical, cognitive, and psychosocial functioning (Minimum value: 0; maximum value: 84; higher scores mean a worse outcome).
Change in the Short Form Health Survey (SF-36) score | Baseline (T0), after 5 days of sports activity (Ti, if applicable), after 8 weeks (T1), after 16 weeks (T2)
  The SF-36 is a patient reported outcome that quantifies health status and measures health-related quality of life (Minimum value: 0%; maximum value: 100%; higher scores mean a better outcome)
Structural and functional plasticity of the Central Nervous System (CNS) | Baseline (T0), after 8 weeks (T1), after 16 weeks (T2)
  Brain structure and function will be investigated using Magnetic Resonance Imaging (MRI) and Transcranial Magnetic Stimulations (TMS) in order to detect possible changes induced by the intervention.
  MRI measures: axial single-shot spin-echo echo-planar diffusion tensor imaging (DTI) to obtain DTI-derived parametric maps (in particular, fractional anisotropy, axial diffusivity, radial diffusivity and mean diffusivity) TMS measures: motor evoked potential of 1mV at rest (S1mV) in the opponens pollicis (OP) before and after paired associative stimulation (PAS), a protocol known to induce a plastic increase of the primary motor cortex (M1) excitability. PAS consists of an electric stimulus delivered on the median nerve of the right arm 25ms (PAS 25) coupled with a magnetic stimulus administered on M1 in correspondence to the OP area. Two-hundred couples of stimuli will be administered to each participants for a total duration of 14 minutes.
Interview | Up to 2 years after the intervention
  Semi-structured interview deputed to explore eventual long-term effects of the intervention and effects on daily living activities and quality of life.
Change in the Hand Grip Strength Test (HGST) performance | Baseline (T0), after 5 days of sports activity (Ti, if applicable), after 8 weeks (T1), after 16 weeks (T2)
  HGST is a tool measuring the maximum isometric strength of the hand and forearm muscles
Change in the Pinch Strength Test (PST) performance | Baseline (T0), after 5 days of sports activity (Ti, if applicable), after 8 weeks (T1), after 16 weeks (T2)
  PST is a tool measuring the maximum isometric strength between thumb and index
Change in the Timed Up and Go (TUG) performance | Baseline (T0), after 5 days of sports activity (Ti, if applicable), after 8 weeks (T1), after 16 weeks (T2)
  TUG is a simple evaluative test used to measure functional mobility
Change in the Timed Up and Go cognitive (TUG-cog) performance | Baseline (T0), after 5 days of sports activity (Ti, if applicable), after 8 weeks (T1), after 16 weeks (T2)
  TUG-cog is a simple evaluative test used to measure functional mobility during dual-task performances
Change in the Arm Function in Multiple Sclerosis Questionnaire (AMSQ) score | Baseline (T0), after 5 days of sports activity (Ti, if applicable), after 8 weeks (T1), after 16 weeks (T2)
  The AMSQ is a patient reported outcome on upper limb functioning (Minimum value: 31; maximum value: 186; higher scores mean a worse outcome)
Change in the 12-Item MS Walking Scale (MSWS-12) score | Baseline (T0), after 5 days of sports activity (Ti, if applicable), after 8 weeks (T1), after 16 weeks (T2)
  MSWS-12 is a self-report measure of the impact of MS on the individual's walking ability (Minimum value: 12; maximum value: 60; higher scores mean a worse outcome).
Change in the Dual-task Impact of Daily Activities Questionnaire (DIDA-Q) score | Baseline (T0), after 5 days of sports activity (Ti, if applicable), after 8 weeks (T1), after 16 weeks (T2)
  DIDA-Q is a self-report measure of the perceived difficulties of dual-tasking (Minimum value: 0; maximum value: 76; higher scores mean a worse outcome)
Change in the Brief Illness Perception Questionnaire (Brief IPQ) score | Baseline (T0), after 5 days of sports activity (Ti, if applicable), after 8 weeks (T1), after 16 weeks (T2)
  Brief IPQ is a self-report measure of illness perceptions (Minimum value: 0; maximum value: 70; higher scores mean a worse outcome)
Continuous monitoring of the time of activity | Baseline (i.e., 1 month before intervention), during sports activity (if applicable) and 1 month after intervention
  A tracker (smart watch or bracelet) monitors the time of activity of participants (minutes/day).
Continuous monitoring of calories expenditure | Baseline (i.e., 1 month before intervention), during sports activity (if applicable) and 1 month after intervention
  A tracker (smart watch or bracelet) monitors the calories expenditure (calories/day).
Questionnaire on acceptability | After 5 days of sports activity (if applicable)
  Yes/No questionnaire composed by five questions evaluating satisfaction the intervention and its organization

CONTACTS AND LOCATIONS:
Overall Officials: Giampaolo Brichetto, MD, PhD, Principal Investigator — Italian Multiple Sclerosis Association and Foundation
Locations (1):
- Italian Multiple Sclerosis Association and Foundation, Genoa, GE, Italy